CLINICAL TRIAL: NCT00292448
Title: A Randomised, Double-blind, Double-dummy, Crossover Efficacy and Safety Comparison of 4-week Treatment Periods of Ba 679 BR Respimat® 5 μg and Tiotropium Inhalation Capsule 18 μg in Patients With COPD
Brief Title: A Randomised, Double-blind, Crossover Study of Ba679BR Respimat in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.291
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Inhalation

INTERVENTIONS:
Drug: Ba 679 BR Respimat
Drug: Tiotropium (Spiriva) inhalation capsule 18 ug

SUMMARY:
The objective of this trial is to compare the efficacy and the safety of Ba 679 BR Respimat 5 ug once daily to tiotropium inhalation capsule 18 ug (Spiriva inhalation capsule) in a crossover study of 4-week treatment periods in patients with COPD.

DETAILED DESCRIPTION:
This is a 16-week, multi-centre, randomised, double-blind, double-dummy, crossover study of 4-week randomised treatment periods to demonstrate the efficacy and safety of 5 ug of Ba 679 BR inhalation solution from Respimat compared to tiotropium inhalation powder capsule (18 ug) via HandiHaler in patients with COPD. The two 4-week randomised treatment periods are separated by 4-week washout period.

Study Hypothesis:

The primary aim of this trial is to demonstrate non-inferiority of lung function response to 5 ug (2 actuations of 2.5 ug) of Ba679BR Respimat delivered by the Respimat inhaler once daily compared to tiotropium (18 ug) inhaled as powder capsule from the HandiHaler once daily at the end of 4-week treatment periods in patients with COPD. The hypothesis test of non-inferiority will be performed at alpha = 0.025 (one-sided).

Comparison(s):

The primary efficacy endpoint is the trough FEV1 response determined at the end of each 4-week period of randomised treatment.

ELIGIBILITY:
participation in the trial 2. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:

? Patients must have relatively stable, moderate to severe airway obstruction with an FEV1 =< 70% of predicted normal* and FEV1 =< 70% of FVC (Visits 1 and 2).

*: Predicted normal values will be calculated according to the formulas for Japanese predicted normal values (R05-0607) (see below).

Males: FEV1 predicted (L) = 0.036 x (height (cm)) ? 0.028 x age (years) ? 1.178 Females: FEV1 predicted (L) = 0.022 x (height (cm)) ? 0.022 x age (years) ? 0.005

? Patients must maintain stable COPD medications for 1 month prior to Visit 1. 3. Male or female patients 40 years of age or older. 4. Patients must be current or ex-smokers with a smoking history of more than 10 pack years.

Pack Years = [Number of cigarettes/ day / 20] x years of smoking 5. Patients must be able to perform technically acceptable pulmonary function tests.

6. Patients must be able to inhale medication in a competent manner from the Respimat inhaler and the HandiHaler.

Patients with/who:

1. Significant diseases except COPD
2. Clinically relevant abnormal haematology, blood chemistry, or urinalysis
3. Recent history of MI
4. Any cardiac arrhythmia requiring drug therapy or who have been hospitalised for heart failure within the past 3 yrs
5. Cancer within the last 5 yrs
6. Symptomatic prostatic hypertrophy or bladder neck obstruction
7. Narrow-angle glaucoma
8. History of asthma, allergic rhinitis, atopic disease, or who have a total blood eosinophil count >= 600 mm3
9. History of life-threatening pulmonary obstruction, or cystic fibrosis or clinically evident bronchiectasis
10. Active tuberculosis
11. History of and/or active significant alcohol or drug abuse
12. Underwent thoracotomy with pulmonary resection
13. Completed a pulmonary rehabilitation program within the 6 weeks prior to the Scr. Visit or who are currently in a pulmonary rehabilitation program
14. Regularly use daytime oxygen for more than 1 h/day and in the investigator?s opinion unable to abstain from the use of oxygen
15. Took an investigational drug within 1 m or 6 half lives prior to Scr. Visit
16. Beta-blockers
17. Anti-allergic drugs or antihistamines for asthma, allergic rhinitis, atopic disease, or other allergic disease with a total blood eosinophil count >= 600 mm3
18. Oral corticosteroids at unstable doses or at doses in excess of the equivalent of 10 mg of prednisone/day or 20 mg every other day
19. Hypersensitivity to anticholinergic drugs, or components of the Respimat delivery system, to lactose or any other component of the inhalation capsule deliver system
20. Pregnant or suspect of pregnant or women who are willing to become pregnant during the study period or nursing women
21. Who are currently participating in another study
22. The randomisation of patients with any respiratory infection or COPD exacerbation in the 6 weeks prior to the Scr. Visit or during the scr. period should be postponed

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157
Dates: Start 2006-02; Study Completion 2007-03

PRIMARY OUTCOMES:
The primary outcome is the trough FEV1 response determined at the end of each 4-week period of randomised treatment.

SECONDARY OUTCOMES:
Trough FVC response after 4 weeks, peak response (FEV1 and FVC) to first dose, peak response (FEV1 and FVC) after 4 weeks, FEV1 AUC0-3h and FVC AUC0-3h response to first dose and after 4 weeks, individual FEV1and FVC measurements at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Nippon Boehringer Ingelheim Co., Ltd.
Locations (25):
- Japan (25):
  - Boehringer Ingelheim Investigational Site, Akita, Akita
  - Boehringer Ingelheim Investigational Site, Bunkyo-ku, Tokyo
  - Boehringer Ingelheim Investigational Site, Bunkyo-ku,Tokyo
  - Boehringer Ingelheim Investigational Site, Habikino, Osaka
  - Boehringer Ingelheim Investigational Site, Inashiki-gun, Ibaraki
  - Boehringer Ingelheim Investigational Site, Itami, Hyogo
  - Boehringer Ingelheim Investigational Site, Kamogawa, Chiba
  - Boehringer Ingelheim Investigational Site, Kishiwada, Osaka
  - Boehringer Ingelheim Investigational Site, Komaki, Aichi
  - Boehringer Ingelheim Investigational Site, Kurume, Fukuoka
  - Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - Boehringer Ingelheim Investigational Site, Matsumoto, Nagano
  - Boehringer Ingelheim Investigational Site, Morioka, Iwate
  - Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - Boehringer Ingelheim Investigational Site, Osakasayama, Osaka
  - Boehringer Ingelheim Investigational Site, Sakai, Osaka
  - Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - Boehringer Ingelheim Investigational Site, Seto, Aichi
  - Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - Boehringer Ingelheim Investigational Site, Takatsuki, Osaka
  - Boehringer Ingelheim Investigational Site, Toyonaka, Osaka
  - Boehringer Ingelheim Investigational Site, Tsukuba, Ibaraki
  - Boehringer Ingelheim Investigational Site, Wakayama, Wakayama
  - Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site, Yokote, Akita